CLINICAL TRIAL: NCT05138289
Title: The REVEALPLAQUE Study: A pRospEctiVe, multicEnter Study to AnaLyze PLAQUE Using CCTA
Acronym: REVEALPLAQUE
Status: Completed | Type: Observational
Sponsor: HeartFlow, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP- 908-001
Record Dates: First submitted 2021-09-24; First posted 2021-11-30 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Disease (CAD) (E.G., Angina, Myocardial Infarction, and Atherosclerotic Heart Disease (ASHD))
MeSH Terms: conditions — Coronary Artery Disease; Angina Pectoris; Myocardial Infarction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Total Plaque Volume — Compare total plaque volume with IVUS obtained during ICA (invasive coronary angiography)

SUMMARY:
This study will evaluate the level of agreement between noninvasive CCTA (coronary computed tomography angiography)-based quantification and characterization of coronary atherosclerosis and invasive IVUS (intravascular ultrasound).

DETAILED DESCRIPTION:
This is a prospective, multi-center study. All patients who have a stenosis in at least one major epicardial vessel confirmed by CCTA, who have undergone FFRCT (Fractional flow reserve-computed tomography) analysis, and who are scheduled to undergo clinically indicated IVUS-guided invasive evaluation and/or treatment will be eligible for enrollment. Enrolling sites will have FFRCT analysis incorporated when indicated into their standard evaluation of CCTA scans. Data collected will include CCTA and FFRCT, full angiographic, and IVUS images, and if obtained, any other imaging or physiologic data including OCT (Optical coherence tomography), FFR (fractional flow reserve), any NHPR (non-hyperemic pressure ratios) (e.g., dPR (diastolic pressure ratio), RFR (resting full-cycle ratio), iFR (instantaneous wave-free ratio), etc.), and pre- and post-stent implantation invasive data. All non-invasive and invasive data collected will be obtained as clinical practice consistent with standard clinical care.

ELIGIBILITY:
Inclusion criteria (all must be present):

1. Age ≥18 years
2. Clinically stable patient with known CAD
3. CCTA showing stenosis in at least one major epicardial vessel of stentable/graftable diameter, in whom clinically indicated IVUS is planned within 45 days of the CCTA and FFRct available
4. FFRct successfully processed
5. Willing to comply with all aspects of the protocol
6. Agrees to be included in the study and able to provide written informed consent.

Exclusion criteria (all must be absent):

1. 1. CCTA showing no stenosis
2. Uninterpretable CCTA by HeartFlow assessment, in which image quality prevents FFRCT from being processed.
3. Acute chest pain
4. CABG (coronary artery bypass graft) prior to CCTA acquisition
5. Prior history of PCI for 3 or more vessels
6. MI (myocardial infarction) less than 30 days prior to CCTA or between CCTA and ICA.
7. Suspicion of acute coronary syndrome (acute myocardial infarction or unstable angina)
8. Known complex congenital heart disease
9. Tachycardia or significant arrhythmia
10. Subject requires an emergent procedure
11. Evidence of ongoing or active clinical instability, including acute chest pain (sudden onset), cardiogenic shock, unstable blood pressure with systolic blood pressure <90 mmHg, and severe congestive heart failure (NYHA [New York Heart Association] III or IV) or acute pulmonary edema
12. Any active, serious, life-threatening disease with a life expectancy of less than 2 months
13. Currently enrolled in another study utilizing FFRCT or in an investigational trial that involves a non-approved cardiac drug or device
14. Persons under the protection of justice, guardianship, or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinically stable patients with known CAD who have a CCTA showing stenosis in at least one major epicardial vessel of stentable/graftable diameter and in whom clinically-indicated IVUS is planned.
Sampling Method: Non-Probability Sample
Enrollment: 258 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jagat Narula, MD, Principal Investigator — HeartFlow Investigative Site; Thomas Stuckey, MD, Principal Investigator — HeartFlow Investigative site; Gaku Nakazawa, MD, Principal Investigator — HeartFlow investigative site
Locations (1):
- HeartFlow Investigative Site, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- IVUS: All patients who have a stenosis in at least one major epicardial vessel confirmed by CCTA, who have undergone FFRCT analysis, and who are scheduled to undergo clinically indicated IVUS-guided invasive evaluation and/or treatment will be eligible for enrollment.
Period: Overall Study
Arm/Group | IVUS
Started | 258
Completed | 258
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Baseline participants is not the same as the Participant flow as 21 participants were excluded from analysis due to technical limitations and we were not able to process medical imaging data.
Arm/Group | IVUS
Number analyzed (Participants) | 237
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61
  Male | 176
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9
  Not Hispanic or Latino | 227
  Unknown or Not Reported | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 157
  Race: Black or African American | 9
  Race: Asian | 63
  Race: American Indian or Alaska Native | 0
  Race: Native Hawaiian or other Pacific Islander | 0
  Race: Other | 8

OUTCOME MEASURES:

1. Primary Outcome: Comparison of Total Plaque Volume
Description: Level of agreement between total plaque volume measured by AI-QCPA (Artificial intelligence quantitative coronary plaque analysis) and IVUS (intravascular ultrasound).
Time Frame: 13 months
Population: as for baseline characteristics
Measure: Number; unit: Pearson's correlation statistic
Arm/Group | IVUS
Number analyzed (Participants) | 237
Pearson's correlation statistic | 0.91

ADVERSE EVENTS:
Time Frame: No adverse event data was collected. This was an observational study and all patients received standard clinical care, no intervention was given.
Description: No adverse event data was collected. This was an observational study and all patients received standard clinical care, no intervention was given. The total number of participants at risk is "0" because there was no adverse event data collected.
Arm/Group | IVUS
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT05138289/Prot_SAP_000.pdf